CLINICAL TRIAL: NCT00019487
Title: Treatment of Patients With Metastatic Melanoma Using Cloned Peripheral Blood Lymphocytes Sensitized In Vitro to the gp209-2M Immunodominant Peptide
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066287; NCI-98-C-0095; NCI-T98-0012; NCT00001694 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2003-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: gp209-2M antigen
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells may make the body build an immune response and kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have metastatic melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether reinfused activated cells alone or in conjunction with high or subcutaneous dose interleukin-2 may result in clinical tumor regression in patients with metastatic melanoma who had previously failed therapy on protocols involving immunization against the gp100 molecule.
* Determine the survival of infused cells with antitumor activity in these patients.

OUTLINE: This is a salvage regimen.

Patients undergo leukopheresis to obtain peripheral blood mononuclear cells or tumor biopsy to obtain tumor infiltrating lymphocytes (TIL). Cells are incubated in the presence of gp209-2M peptide and then harvested and cloned. Patients receive 30-minute IV infusions of these in vitro sensitized cells. Treatment repeats every 2 weeks for 2 courses. An additional cohort of 8 patients receives gp209-2M peptide in Montanide ISA-51 subcutaneously in 2 different sites followed 2 days later by the adoptive transfer of cloned lymphocytes. At 4 to 6 weeks after the treatment courses, patients with stable or regressing disease may be retreated.

Patients with disease progression after 2 courses may receive 2 additional courses of cell infusion followed by interleukin-2 (IL-2) on one of two schedules. One cohort of patients receives IL-2 by intravenous bolus over 15 minutes every 8 hours beginning on the day after cell infusion and continuing for up to 5 days of each treatment course. Another cohort receives IL-2 by daily subcutaneous injections on days 1-12 of each course of therapy. If after 12-16 patients have been treated with cloned cells alone initially and responses are inadequate, subsequent patients entered into this study are randomized to receive the cell infusion followed by IL-2 on one of the two described schedules.

Patients are followed at 4-6 weeks.

PROJECTED ACCRUAL: A total of 91 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic melanoma that has failed therapy on protocols involving immunization against the gp100 molecule
* Measurable or evaluable metastatic disease
* Must be HLA-A201 positive by standard HLA typing

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 3 months

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.0 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT/AST less than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.6 mg/dL

Cardiovascular:

* For patients randomized to receive interleukin-2:

  * No major medical illnesses of the cardiovascular system

Pulmonary:

* For patients randomized to receive interleukin-2:

  * No major medical illnesses of the pulmonary system

Other:

* HIV negative
* Hepatitis B antigen negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* For patients randomized to receive interleukin-2:

  * No active systemic infection
  * No other major medical illnesses of immune system
  * No coagulation disorders

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* No concurrent steroid therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No concurrent active treatment of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dudley ME, Wunderlich J, Nishimura MI, Yu D, Yang JC, Topalian SL, Schwartzentruber DJ, Hwu P, Marincola FM, Sherry R, Leitman SF, Rosenberg SA. Adoptive transfer of cloned melanoma-reactive T lymphocytes for the treatment of patients with metastatic melanoma. J Immunother. 2001 Jul-Aug;24(4):363-73. doi: 10.1097/00002371-200107000-00012. PMID 11565838